CLINICAL TRIAL: NCT02372305
Title: Comparison of FlexHD and Alloderm Outcomes in Breast Reconstructive Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI is no longer at institution. IRB closed study due to lack of response from PI
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 203456
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — FlexHD; Alloderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FlexHD (Active Comparator): Patients randomly assigned to receive FlexHD for breast reconstruction.
  Interventions: Biological: FlexHD
- Alloderm (Active Comparator): Patients randomly assigned to receive Alloderm for breast reconstruction.
  Interventions: Biological: Alloderm

INTERVENTIONS:
Biological: FlexHD — Patients will be randomized to receive FlexHD.
  Arms: FlexHD
Biological: Alloderm — Patient will be randomized to receive Alloderm.
  Arms: Alloderm

SUMMARY:
FlexHD and Alloderm are two common products used in breast reconstruction to hold tissue expanders and implants in place. There have been few chart review studies comparing outcomes between the two materials in breast reconstruction. These studies have determined there is no difference in complication rates between the two materials. However, there have never been any active studies to date. This study will serve as a randomized controlled trial comparing FlexHD and Alloderm. Several outcomes will be measured based off of inclusion and exclusion criteria to determine if either product is more suitable for use in breast reconstruction. This will be performed by randomly assigning patients to receive either FlexHD or Alloderm. Designated outcomes will be followed closely postoperatively. Outcomes will be statistically analyzed to determine complication rates between FlexHD and Alloderm and thus which product is better to use in breast reconstruction.

DETAILED DESCRIPTION:
FlexHD and Alloderm are two common products used in breast reconstruction to hold tissue expanders and implants in place. There have been few chart review studies comparing outcomes between the two materials in breast reconstruction. These studies have determined there is no difference in complication rates between the two materials. However, there have never been any active studies to date. This study will serve as a randomized controlled trial comparing FlexHD and Alloderm. Several outcomes will be measured based off of inclusion and exclusion criteria to determine if either product is more suitable for use in breast reconstruction. This will be performed by randomly assigning patients to receive either FlexHD or Alloderm. Designated outcomes will be followed closely postoperatively. Outcomes will be statistically analyzed to determine complication rates between FlexHD and Alloderm and thus which product is better to use in breast reconstruction

ELIGIBILITY:
Inclusion Criteria:

* BMI<30
* No Prior Breast Radiation
* No Prior Breast Reduction
* No Diabetes Mellitus (IDDM and non-IDDM)
* Non-smoker or quit >6 weeks prior
* No breast implants or prior breast implants
* No inflammatory or autoimmune disorders
* No current anticoagulation therapy
* No current pregnant

Exclusion Criteria:

* BMI > 30
* Prior Breast Radiation
* Diabetes Mellitus - IDDM and non IDDM
* Prior Breast Reduction
* Active Smoker or Recently Quit <6 weeks
* Prior Breast Implants
* Inflammatory/Autoimmune Condition (ex. Lupus)
* Current Anticoagulation Therapy
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Wound Dehiscence | One Year
  time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Pallavi A Kumbla, MD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yuen JC, Yue CJ, Erickson SW, Cooper S, Boneti C, Henry-Tillman R, Klimberg S. Comparison between Freeze-dried and Ready-to-use AlloDerm in Alloplastic Breast Reconstruction. Plast Reconstr Surg Glob Open. 2014 Apr 7;2(3):e119. doi: 10.1097/GOX.0000000000000061. eCollection 2014 Mar. PMID 25289313
- [Background] Liu DZ, Mathes DW, Neligan PC, Said HK, Louie O. Comparison of outcomes using AlloDerm versus FlexHD for implant-based breast reconstruction. Ann Plast Surg. 2014 May;72(5):503-7. doi: 10.1097/SAP.0b013e318268a87c. PMID 23636114
- [Background] Brooke S, Mesa J, Uluer M, Michelotti B, Moyer K, Neves RI, Mackay D, Potochny J. Complications in tissue expander breast reconstruction: a comparison of AlloDerm, DermaMatrix, and FlexHD acellular inferior pole dermal slings. Ann Plast Surg. 2012 Oct;69(4):347-9. doi: 10.1097/SAP.0b013e31824b3d97. PMID 22868313